CLINICAL TRIAL: NCT06737510
Title: Improving Emergency Preparedness Among 9/11 Exposed Population: Implementation and
Brief Title: Improving Emergency Preparedness Among 9/11 Exposed Population: Implementation and Evaluation of an Emergency Preparedness Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York City Department of Health and Mental Hygiene (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-150
Record Dates: First submitted 2024-10-09; First posted 2024-12-17 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Emergency Preparedness

STUDY DESIGN:
Intervention Model Description: A two-arm parallel randomized controlled trial will be conducted to compare the effectiveness of a phone-based household emergency preparedness intervention with a mailed informational brochure on household emergency preparedness amongst a sample of World Trade Center Health Registry enrollees residing within New York City.
Masking Description: N/A No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phone-based household emergency preparedness (Experimental): A phone-based intervention will consist of 15 - 20 minutes discussion covering the following topics: (1) an introduction to why emergency preparedness is important; (2) definition of what a disaster is; (3) family communication plan (including, what is a family communication and evacuation plan, why you should have one, communication plan checklist, including a family communication card); (4) disaster supplies (including, what types of supplies are needed, how long supplies should last, supply checklist, and storing supplies); and (5) resources (including providing NYC Emergency Management website: NYC.gov/hazards, i which includes specific information related to the participants New York City hurricane evacuation zones) .
  Interventions: Behavioral: Phone-based household emergency preparedness
- Informational brochure on household emergency preparedness (Experimental): An informational brochure will be mailed to participants and will cover the following topics: (1) an introduction to why emergency preparedness is important; (2) definition of what a disaster is; (3) family communication plan (including, what is a family communication and evacuation plan, why you should have one, communication plan checklist, family communication card); (4) disaster supplies (including, what types of supplies are needed, how long supplies should last, supply checklist, and storing supplies, including preparing a go bag); and (5) resources (including disaster contact numbers for emergency and non-emergency calls (911 and 311), how to register for emergency notifications ("Notify NCY"), NYC Emergency Management, as well as a website for additional information on preparedness (NYC.gov/hazards) that includes New York City hurricane evacuation zones .
  Interventions: Behavioral: Informational brochure on household emergency preparedness

INTERVENTIONS:
Behavioral: Informational brochure on household emergency preparedness — An informational brochure will be mailed to participants and will cover the following topics: (1) an introduction to why emergency preparedness is important; (2) definition of what a disaster is; (3) family communication plan (including, what is a family communication and evacuation plan, why you should have one, communication plan checklist, family communication card); (4) disaster supplies (including, what types of supplies are needed, how long supplies should last, supply checklist, and storing supplies, including preparing a go bag); and (5) resources (including disaster contact numbers for emergency and non-emergency calls (911 and 311), how to register for emergency notifications ("Notify NCY"), NYC Emergency Management, as well as a website for additional information on preparedness (NYC.gov/hazards) that includes New York City hurricane evacuation zones .
  Arms: Informational brochure on household emergency preparedness
Behavioral: Phone-based household emergency preparedness — A phone-based intervention will consist of 15 - 20 minutes discussion covering the following topics: (1) an introduction to why emergency preparedness is important; (2) definition of what a disaster is; (3) family communication plan (including, what is a family communication and evacuation plan, why you should have one, communication plan checklist, including a family communication card); (4) disaster supplies (including, what types of supplies are needed, how long supplies should last, supply checklist, and storing supplies); and (5) resources (including providing NYC Emergency Management website: NYC.gov/hazards, i which includes specific information related to the participants New York City hurricane evacuation zones) .
  Arms: Phone-based household emergency preparedness

SUMMARY:
A two-arm parallel randomized controlled trial will be conducted to compare the effectiveness of a phone-based household emergency preparedness intervention with a mailed informational brochure on household emergency preparedness amongst a sample of World Trade Center Health Registry enrollees residing within New York City.

DETAILED DESCRIPTION:
An intervention to enhance household emergency preparedness was developed to include the following topics: (1) an introduction to why emergency preparedness is important; (2) definition of what a disaster is; (3) family communication and evacuation plan (including, what is a family communication plan, why you should have one, communication plan checklist, family communication card); (4) disaster supplies (including, what types of supplies are needed, how long supplies should last, supply checklist; assembling a go bag , and storing supplies); and (5) The brochure included several resources, including disaster contact numbers for emergency and non-emergency calls: 911 or 311,, NYC Emergency Management, as well as website for additional information of preparedness: NYC.gov/hazards, which includes information specific to New York City hurricane evacuation zones.

The phone-based intervention consisted of a 15 - 20 minutes talk session completed over the phone following the format and topics noted above. The informational brochure intervention followed the format and topic above and was mailed to participants during the intervention period.

ELIGIBILITY:
Inclusion Criteria:

1. English or Spanish speaking World Trade Center Health Registry enrollees aged 18 or older at the time of 9/11 residing in New York City.
2. Completed Wave 4 (2015-2016)
3. Those who are not rescue/recovery workers in either the NYPD or FDNY.

   -

Exclusion Criteria:

1. World Trade Center Health Registry enrollees under the age of 18 at the time of 9/11
2. Those with proxy interview at Wave 1
3. Enrollee was a rescue and recovery work affiliated with FDNY or NYPD at Wave 1

   -

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 707 (Estimated)
Dates: Start 2018-11-21 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
The CASPER instrument sum score | up to 24 weeks
  The primary outcome is based on the CDC CASPER emergency preparedness instrument. It consists of ten yes/no questions, five relating to having a communication plan and five related to having an emergency supply kit. The primary outcome is the sum of the number of questions answered "yes" by the subject.

SECONDARY OUTCOMES:
Individual CASPER instrument items | up to 24 weeks
  Secondary outcomes will be each of the ten individual yes/no questions of the CASPER instrument.

CONTACTS AND LOCATIONS:
Locations (1):
- NYCDOHMH, New York, New York, United States